CLINICAL TRIAL: NCT01738347
Title: Assess Safety, Bio-distribution, and Radiation Dosimetry, and Optimize the Imaging Protocol of GEH120714 (18F) Injection, a Marker of Microglial Activation, in Healthy Volunteers and Participants With Relapsing and Remitting Multiple Sclerosis (rrMS)
Brief Title: Assess Safety, Bio-distribution, Radiation Dosimetry and Optimize the Imaging Protocol of GEH120714 (18F) Injection in Healthy Volunteers and Participants With Relapsing and Remitting Multiple Sclerosis (rrMS).
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GE Healthcare (Industry)
Collaborators: Centre for Probe Development and Commercialization (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: GE-180-001
Record Dates: First submitted 2012-11-13; First posted 2012-11-30 (Estimated); Last update posted 2017-02-24 (Actual); Status verified 2017-02

CONDITIONS: Relapsing-remitting Multiple Sclerosis (rrMS)
MeSH Terms: conditions — Multiple Sclerosis, Relapsing-Remitting | interventions — Injections

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Arm 1 - GEH120714 (18F) Injection (Experimental): Intervention is to administer GEH120714 (18F) Injection (100-270 Megabecquerel (MBq), single intravenous administration).
  Interventions: Drug: Arm 1 - GEH120714 (18F) Injection

INTERVENTIONS:
Drug: Arm 1 - GEH120714 (18F) Injection — Intervention is to administer GEH120714 (18F) Injection (100-270 Megabecquerel (MBq), single intravenous administration).
  Other Names: GEH120714 (18F)

SUMMARY:
To evaluate the safety, bio-distribution, and radiation dosimetry; and to optimize the Imaging Protocol of GEH120714 (18F) Injection. Study recruits healthy volunteers and participants with relapsing and remitting multiple sclerosis.

ELIGIBILITY:
Inclusion Criteria:

Inclusion Criteria for all Participants:

* The subject has a clinically normal or acceptable medical history and physical examination at screening.
* The subject has an acceptable kidney function (eGFR >60 mL/min/1.73m2) for administration of Gadolinium.
* The subject has a trans-locator protein (TSPO) platelet assay conducted with documented results.

Inclusion Criteria for all healthy volunteers:

* The subject has no clinical history or signs of neurological impairment.
* The subject has a normal MRI without central white white matter lesions.

Inclusion Criteria specific for participants with relapsing and remitting results sclerosis (rrMS):

* Subject with a previous diagnosis of rrMS, presenting with (a) clinically active disease at time of screening or, or preferentially, (b) clinically active disease at time of screening and having at least one gadolinium--enhanced lesion on MRI.
* The subject at screening has a MRI scan of sufficient quality for Volume of Interest (VOI) definition and co-alignment with Positron Emission Tomography (PET).

Exclusion Criteria:

General Exclusion Criteria for all participants:

* The subject has a contraindication for Magnetic Resonance Imaging (MRI).
* The subject has known allergies to Gadolinium contrast agent.
* The subject has received significant ionising radiation exposure from clinical trials or medical examinations in the last 12 months.

Exclusion Criteria specific for healthy volunteers:

* The subject has family history of multiple sclerosis (MS).
* The subject is undergoing monitoring of occupational ionising radiation exposure.

Exclusion Criteria specific for participants with remitting multiple sclerosis (rrMS):

* The subject has a past history of cerebrovascular disease or vasculitis.
* The subject has a history of head injury with prolonged coma.

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2013-04; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Recording the occurrence of adverse events (AEs) to evaluate the safety of a single dose of GEH120714 (18F) Injection in healthy volunteers (HV) and participants with rrMS. | Time zero equals the date of contrast imaging and for up to 24 hours for safety monitoring post contrast administration.
  Record the occurrence of adverse events (AEs) to evaluate the safety of a single dose of GEH120714 (18F) Injection in healthy volunteers (HV) and participants with rrMS.

SECONDARY OUTCOMES:
Blood samples collected multiple periods post injection; and urine samples at periods post injection to count radioactivity to determine bio-distribution, internal radiation dosimetry and Effective Dose (E) in healthy volunteers (HV). | Time zero equals the date of contrast imaging and up to the evaluation of the images and the kinetic modelling of cerebral uptake of GEH120714 (18F) Injection,
  Collect blood samples at multiple time periods up to 120 minutes post drug injection; and urine samples at multiple time periods up to 270 minutes post drug injection to count radioactivity to determine the bio-distribution, internal radiation dosimetry and Effective Dose (E) per protocol in healthy volunteers (HV).

CONTACTS AND LOCATIONS:
Overall Officials: Paul Sherwin, M.D., Study Director — GE Healthcare
Locations (1):
- St. Joseph Healthcare, Hamilton, Ontario, Canada